CLINICAL TRIAL: NCT02655705
Title: Comparison of the Performance of Subjective or Objective Psoriasis Severity Assessment Tools for the Assessment of the Improvement of Psoriasis After Oral Cyclosporine A or Methotrexate Treatment
Brief Title: Comparison Study of Psoriasis Severity Assessment Tools
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Woong Youn, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oPASI1403
Record Dates: First submitted 2016-01-04; First posted 2016-01-14 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Psoriasis
Keywords: Cyclosporine; Methotrexate
MeSH Terms: conditions — Psoriasis | interventions — Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine A (Active Comparator): Cyclosporine 200 mg/day (male) and 150 mg/day (female) orally, divided twice daily for 16 weeks
  Interventions: Drug: Cyclosporine A
- Methotrexate (Active Comparator): Methotrexate was started with 10 mg/week orally as a single dose, increasing 2.5 mg every 2 weeks up to 15 mg/week maintenance dose
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Cyclosporine A — Male 200 mg/day, Female 150 mg/day for 16 weeks
  Other Names: Cyclosporin; Ciclosporin; Cyclosporin A
  Arms: Cyclosporine A
Drug: Methotrexate — Initial dose with 10 mg/week, increasing 2.5 mg every 2 weeks up to 15 mg/week maintenance dose
  Other Names: Methotrexate tab
  Arms: Methotrexate

SUMMARY:
This study evaluates the performance of objective psoriasis severity assessment tool compared with a subjective assessment tool for the assessment of the improvement of psoriasis after oral cyclosporine A or methotrexate treatment.

DETAILED DESCRIPTION:
Patients with moderate-to-severe psoriasis were randomly assigned to treatment for 16 weeks with either cyclosporine A (20 patients; male 200 mg/day, female 150 mg/day) or methotrexate (20 patients; initial dose with 10 mg/week, increased up to 15 mg/week). The primary outcome was to compare the difference between the conventional subjective Psoriasis Area and Severity Index (PASI) and the objective PASI by using Colorimeter at 2, 4, 8, 12, and 16 weeks of treatment. The secondary outcome was differences between cyclosporine and methotrexate for treatment of psoriasis, evaluating clinical efficacy and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic plaque psoriasis based on a clinical diagnosis
* Have > 5% body surface area involvement at screening
* Are a candidate for systemic therapy
* Are male or female patients 18 years or older
* Have given written informed consent approved by the Institutional Review Board

Exclusion Criteria:

* Have predominant pattern of pustular, erythrodermic, or guttate forms of psoriasis
* Have had any of the systemic non-biologic psoriasis therapy (including neotigason, cyclosporine, and methotrexate) within 4 weeks prior to baseline
* Have had etanercept within 4 weeks prior to baseline
* Have had adalimumab and infliximab within 8 weeks prior to baseline
* Have had ustekinumab within 16 weeks prior to baseline
* Presence of significant hepatic or renal disorders
* Have uncontrolled arterial hypertension
* Are women who are lactating, breastfeeding or planning pregnancy
* Have any other condition that precludes from following and completing the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) and Objective PASI (oPASI) change over time | up to 16 weeks
  PASI scores and oPASI scores are carried out on every visit. One dermatologist rates a PASI score. A oPASI score is obtained from oPASI formula using Colorimeter parameters L*, a* and b* values.
  oPASI = 0.1×oPSI (head)×Area (head) + 0.3×oPSI (trunk)×Area (trunk) +0.2×oPSI (arm)×Area (arm) + 0.4×oPSI (leg)×Area (leg)
  oPSI = 0.05 x L* - 2.5 x tan-1 (b*/a*) + 5
  PASI range is 0 to 72 score. oPSI range is 1.073 to 10 score.

SECONDARY OUTCOMES:
Number of participants with abnormal laboratory values and/or adverse events that are related to treatment | Screening, 4, and 12 weeks
  Laboratory tests are performed at screening, 4, and 12 weeks. Patients are checked hemoglobin, hematocrit, white blood cell, platelet, aspartate aminotransferase, alanine aminotransferase, blood urea nitrogen, creatinine, c-reactive protein, and erythrocyte sedimentation. All patients are asked treatment-related adverse events on every visit.
Proportion of patients achieving 75% and 90% PASI improvement on every visit | up to 16 weeks
  Investigators evaluate proportions of patients showing at least 75% and 90% improvement from baseline in PASI.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Woong Youn, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available within 6 months of study completion.

REFERENCES:
- [Background] Choi JW, Kim BR, Choi CW, Youn SW. One device, one equation: the simplest way to objectively evaluate psoriasis severity. J Dermatol. 2015 Feb;42(2):154-8. doi: 10.1111/1346-8138.12727. Epub 2014 Dec 10. PMID 25492025
- [Background] Choi JW, Kwon SH, Youn JI, Youn SW. Objective measurements of erythema, elasticity and scale could overcome the inter- and intra-observer variations of subjective evaluations for psoriasis severity. Eur J Dermatol. 2013 Apr 1;23(2):224-9. doi: 10.1684/ejd.2013.1931. PMID 23518409